CLINICAL TRIAL: NCT03420508
Title: A Phase 2 Study of the ALK Inhibitor Ensartinib for Patients With Melanomas Harboring ALK Alterations or Aberrant ALK Expression
Brief Title: Treating Patients With Melanoma and ALK Alterations With Ensartinib
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Xcovery Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-471
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Melanoma
Keywords: Ensartinib; ALK Inhibitor; ALK Alterations; Aberrant ALK Expression; 17-471
MeSH Terms: conditions — Melanoma | interventions — ensartinib

STUDY DESIGN:
Intervention Model Description: This single arm, single center, open label Phase 2 trial will utilize a Simon 2 stage design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ensartinib (Experimental): The screening portion of the trial will test archival tumor material for the presence of ALKATI using a Nanostring-based RNA assay for any patients deemed to be current or future candidates for this trial. This will require approximately 5 formalin-fixed paraffin- embedded (FFPE) slides of 5-8 micron thickness. For the treatment portion of the study, all patients will receive ensartinib orally at a dose of 225mg daily.
  Interventions: Drug: Ensartinib; Diagnostic Test: ALKATI by Customized Nanostring Assay

INTERVENTIONS:
Drug: Ensartinib — Ensartinib will be given at a dose of 225mg daily in the form of 100mg and 25mg capsules. Patients will receive treatment continuously in 28 day cycles. Patients will then have the same tumor specimen biopsied again at day 15. Treatment will continue until disease progression, unacceptable toxicity, or patient choice to discontinue therapy.
Diagnostic Test: ALKATI by Customized Nanostring Assay — a custom chip with probes targeting the ATI site in ALK, providing a reproducible, quantitative measure of ALKATI

SUMMARY:
The purpose of this study is to test the effects of the study drug, ensartinib, on the patient and the cancer. Ensartinib is a new, investigational type of treatment for melanoma with a particular type of abnormality.

ELIGIBILITY:
Inclusion Criteria:

For Screening Phase:

* Patients ≥18 years of age
* Histologically confirmed advanced malignant melanoma, regardless of subtype

For Treatment Phase, as above and in addition:

* Progression following PD-1 based checkpoint inhibitor therapy, with or without ipilimumab. Tumors harboring BRAF V600 alterations must also have received prior therapy with BRAF inhibitors (with or without a MEK inhibitor). Patients with uveal melanoma are exempt from PD-1 based progression since there is no accepted standard frontline therapy.
* Tumors must harbor an alteration in ALK using a CLIA-certified laboratory, including, but not limited to, ALKATI, ALK fusions, or ALK mutations.
* Disease must be measurable according to RECIST 1.1. Disease that has undergone local therapy in the past 30 days is not considered measurable unless the investigator has documented progression despite the local therapy.

  ° If a patient has consented to the pre-screening portion, has been determined to have ALK alterations, but has no measurable disease, the trial may be favored later, and the patient should be consented (or re-consented) to the treatment portion of the trial at the discretion of the investigator.
* Asymptomatic untreated brain metastases are allowed. Symptomatic metastases that have undergone local therapy with RT or surgery and have not required an increase in steroid dose in prior 2 weeks are allowed. Disease that has undergone local therapy is not considered measurable.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-2
* Acceptable liver, renal, and hematological function:

  * total bilirubin ≤1.5x upper limit of normal (ULN); patients with Gilbert's Syndrome must have bilirubin ≤3x ULN
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤3 x ULN (≤5x if liver metastases are present)
  * Estimated glomerular filtration rate (GFR) ≥ 30 mL/min using a cancer-specific GFR Model; the calculator found at: http://tavarelab.cruk.cam.ac.uk/JanowitzWilliamsGFR/
  * Hemoglobin ≥9 g/dL
  * Neutrophils ≥1.5 x 10^9/L
  * Platelets ≥100 x 10^9/L
  * Prothrombin time, international normalized ratio [INR], and/or activated partial thromboplastin time within ≤1.5 x ULN
* Prothrombin time, international normalized ratio [INR], and/or activated partial thromboplastin time within ≤1.5 x ULN

Exclusion Criteria:

For Screening Phase:

* Any prior ALK inhibition.

For Treatment Phase, as above and in addition:

Prior therapy with immune-activating agents within less than 1 cycle length prior to first day of study treatment (e.g. 3 weeks for ipilimumab or pembrolizumab; 2 weeks for nivolumab).

* Prior therapy with BRAF/MEK agents within 3 weeks prior to first day of study treatment.
* Any other systemic or regional anticancer therapy (cytotoxic chemotherapy, embolization) within 3 weeks or 1 cycle length, whichever is shorter, prior to first day of study treatment
* Prior RT or clinically relevant major surgery (e.g. craniotomy, metastasectomy) within 2 weeks prior to first day of study treatment.
* Any other active malignancy other than melanoma that, in the opinion of the investigator, would interfere with study participation.
* Receipt of any other systemic anticancer therapy except for hormonal therapy for a hormonally sensitive (e.g. breast or prostate) cancer.
* Receipt of strong CYP3A inhibitors or inducers per Appendix A.
* Clinically significant cardiovascular disease, including:

  * QTc interval by Bazett's formula >480 ms
  * Symptomatic bradycardia <45 beats per minute
  * Other clinically significant ECG abnormalities (e.g. bundle branch block) may be eligible after discussion with the Principal Investigator
  * Clinically uncontrolled hypertension in the investigator's opinion.
* The following within 6 months prior to Cycle 1 Day 1:

  * Congestive heart failure (New York Heart Class III or IV).
  * Cardiomyopathy.
  * o Arrhythmia or conduction abnormality requiring medication. Note: patients with atrial fibrillation/flutter adequately controlled by medication in the opinion of the treating physician and arrhythmias controlled by pacemakers are eligible.
  * Severe/unstable angina, coronary artery/peripheral bypass graft, or myocardial infarction.
  * Cerebrovascular accident or transient ischemia.
* Any serious, active infection at the time of treatment such as bacteremia
* Interstitial lung disease or pneumonitis that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity. Patients with prior pneumonitis that has resolved are eligible.
* Patients must not be pregnant or breast feeding, or unable or unwilling to use proper contraception during the study and up to 3 months following study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
clinical benefit rate (CBR) | up to 24 weeks
  CBR is defined as any confirmed objective response by Response Evaluation in Solid Tumor (RECIST) 1.1, or stable disease until the 24 week assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shoushtari, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm